CLINICAL TRIAL: NCT06948838
Title: Comparative Effectiveness of Interventions to Improve Hypertension Control in Safety-Net Settings: The Boston Hypertension Equity Alliance in Treatment
Brief Title: Improving Hypertension Control in Safety-Net Settings: The Boston Hypertension Equity Alliance in Treatment
Acronym: BHEAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Boston Healthcare for the Homeless Program (BHCHP) (Unknown); Boston Medical Center General Internal Medicine primary care (BMC GIM) (Unknown); Boston Medical Center Family Medicine Primary Care (BMC FM) (Unknown); NeighborHealth Center Family Medicine at Maverick Street (NH FM) (Unknown); NeighborHealth Center Internal Medicine at Gove Street (NH IM) (Unknown); NeighborHealth South End (NH South End) (Unknown); Manet Community Health Center (Maner CHC) (Unknown); Mattapan Community Health Center (Mattapan) (Unknown); Greater Roslindale Medical and Dental Center (GRMDC) (Unknown); Boston University School of Public Health (BUSPH) (Unknown); BUSPH Biostatistics and Epidemiology Data Analytics Center (BEDAC) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: H-45398; HMC-2023C2-33345 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2025-04-15; First posted 2025-04-29 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Hypertension; Hypertension Complicated
Keywords: Remote blood pressure monitoring (RBPM); HTN management; HTN-related outcomes; Evidence-based health system strategies; Hybrid effectiveness-implementation study; PROs; Diverse urban area; Disparities
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: A hybrid type 1 effectiveness-implementation study with a cluster randomized stepped wedge study design will be used. This will be a longitudinal repeated measures design. RBPM will begin for all clusters in September, 2025. At the end of month 12, MII implementation will begin for the group in the first wedge, with the second and third groups implementing at 6-month intervals thereafter. All sites will continue interventions as part of ongoing operations, with final long-term follow-up assessment at the end of month 54.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Blood Pressure Monitoring (RBPM) (Experimental): Individual level interventions fo monitor blood pressure.
  Interventions: Behavioral: RBPM
- Multilevel Intensification interventions (MII) (Experimental): Team-based interventions to mitigate clinical inertia which is the lack of intensification of treatment despite inadequate disease control such as for HTN.
  Interventions: Behavioral: RBPM; Other: MII

INTERVENTIONS:
Behavioral: RBPM — Standardized blood pressure measurement and treatment protocols in clinical practice.
Other: MII — Team-based interventions including multiple evidence-proven interventions such as clinician decision support, monitoring medication non-adherence, use of combination pills, and formulary modifications.
  Arms: Multilevel Intensification interventions (MII)

SUMMARY:
High blood pressure (BP) or hypertension (HTN) affects over 100 million individuals in the US, increasing the risk of adverse outcomes, including stroke, myocardial infarction (MI), and chronic kidney disease (CKD). Effective therapies include non-pharmacologic approaches and multiple medication classes. Successful HTN management requires ongoing patient engagement for BP monitoring and treatment intensification. Reaching this goal is challenging, and many patients with HTN do not have controlled BP.

Using a collaborative partnership between patients, clinicians, health system and public health stakeholders, and the research team the investigators plan to overcome barriers to widespread implementation of evidence-based health system strategies to improve BP control in a large, urban, primary care-based safety-net setting for diverse populations experiencing disparities in HTN-related outcomes.

DETAILED DESCRIPTION:
A hybrid type 1 effectiveness-implementation study will be implemented to evaluate the comparative impact of each intervention on clinical outcomes while also assessing implementation at each site. The multi-site cluster randomized stepped-wedge design allows for feasible resource allocation and sequential roll out of the interventions for comparison, ensuring each site has the opportunity to benefit from both approaches. Data will be collected for multiple patient reported outcomes (PROs) to understand the range of impacts of the interventions from the patient perspective.

The specific aims are to:

* Assess comparative effectiveness of remote BP monitoring (RBPM) versus RBPM + multilevel intensification intervention (MII) on HTN control and quality of care. Prior research has demonstrated the effectiveness of each of these interventions yet the optimal approach to achieve equity in HTN control in safety net practices remains unknown.
* Use mixed methods, guided by the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework, to assess implementation of the two comparators as measured by reach, adoption, implementation (fidelity) and maintenance. Using a convergent parallel design, the investigators will use concurrent quantitative and qualitative data to obtain perspectives across multiple levels to understand the reasons for success or failure of implementation of each comparator. By merging these data, integration can be achieved by using qualitative themes related to implementation to support or refute quantitative findings of reach and fidelity.
* Evaluate the comparative impacts of each intervention on PROs assessed with validated measures of patient activation, medication adherence, and trust in medical settings. The study intervention approaches were informed by direct feedback from the targeted diverse patients and clinical providers to address patient-reported barriers to HTN control: lack of activation, adherence to medications, and trust in their care providers.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age>18) patients receiving primary care at one of the 9 participating sites, with primary care provider (PCP) visit in the preceding year
* Presence of HTN defined by one or more of: 1) diagnosis included on active problem list, 2) active HTN medications in prior year, 3) 3 separate elevated BP measurements
* Uncontrolled HTN defined as systolic blood pressure (SBP)>140

Exclusion Criteria:

* Not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16895 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure (SBP) improvement | Baseline, every 3 months up to 54 months
  Change in BP abstracted from the electronic health record (EHR).
Interventions received | Baseline, 54 months
  The number and proportion of individuals who receive each intervention.
Patient activation | Baseline, 18 months, 30 months, 36 months, 42 months, 54 months
  Patient activation will be assessed with the Consumer Health Activation index (CHAI), a 10 item validated instrument that generates a score of 0-100, with ≥80 indicating moderate/high activation.

SECONDARY OUTCOMES:
Blood pressure control | Baseline, 18 months, 30 months, 36 months, 42 months, 54 months
  Assessed as Yes/No from EHR records for Systolic BP<140 mmHg and Systolic BP<130 mmHg.
Medication intensification | Baseline, 18 months, 30 months, 36 months, 42 months, 54 months
  Assessed from EHR and claims data.
BP monitoring | Baseline, 18 months, 30 months, 36 months, 42 months, 54 months
  Assessed by EHR data on the frequency of BP monitoring.
Fidelity of interventions | Baseline, 18 months, 30 months, 36 months, 42 months, 54 months
  The number and proportion of individuals who receive all key elements of the interventions based on EHR data.
Medication adherence | Baseline, 18 months, 30 months, 36 months, 42 months, 54 months
  the 3-item self-report scale by Wilson will be used to assess this outcome. It queries patients about how many days they missed medications and overall consistency over the last 30 days. This measure has been standardized to a 0-100 scale, with good adherence defined as ≥80.
Trust in primary care | Baseline, 18 months, 30 months, 36 months, 42 months, 54 months
  Assessed with the 10 item Wake Forest Physician Trust Scale. The scale uses a 5-point Likert scale [1=strongly disagree to 5=strongly agree]. Total scores can range from 10 to 50, and higher scores represent greater trust.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fischer, MD MS, Principal Investigator — Boston Medical Center, Internal Medicine; Cheryl Clark, MD ScD, Principal Investigator — Institute for Health Equity Research, Evaluation & Policy, MA League of CHCs
Locations (7):
- United States (7):
  - Boston Healthcare for the Homeless (BHCHP), Boston, Massachusetts
  - Boston Medical Center Family Medicine, Boston, Massachusetts
  - Boston Medical Center, General Internal Medicine primary care, Boston, Massachusetts
  - Neighborhood Health, Boston, Massachusetts
  - Mattapan Community Health Center, Boston, Massachusetts
  - Manet Community Health Center, Quincy, Massachusetts
  - Greater Roslindale Medical and Dental Center (GRMDC), Roslindale, Massachusetts

IPD SHARING:
Plan to Share IPD: No